CLINICAL TRIAL: NCT04550091
Title: Role Of Multi-detector Computed Tomography In Differentiation Between Different Types Of Ascites
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Merna youssef nemr, Resident, Assiut University
Other Study IDs: Hounsfields units
Record Dates: First submitted 2020-08-20; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Detection of ascites using CT — Role Of Multi-detector Computed Tomography In Differentiation Between Different Types Of Ascites

SUMMARY:
Role Of Multi-detector Computed Tomography In Differentiation Between Different Types Of Ascites

DETAILED DESCRIPTION:
1. To detect accuracy of MDCT in differentiation between different types of ascites and its underlying cause .
2. To evaluate the diagnostic accuracy of measuring the CT density of the ascitic fluid (in Housefield units) to differentiate between different types of ascites in comparison to aspiration cytology results.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are diagnosed with ascites by clinical examination or by any other investigations such as ultrasound.

Exclusion Criteria:

* Patient with bleeding tendancy and on anticoagulant drugs.-
* Patients who are pregnant .

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are diagnosed with ascites by clinical examination or by any other investigations such as ultrasound.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2020-10-19 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
differentiate between different types of ascites and its underlying cause | 2022
  differentiate between different types of ascites and its underlying causes by measuring the CT density of the ascitic fluid (in Hounsfield units)